CLINICAL TRIAL: NCT07394842
Title: Longitudinal Effects of Head and Neck Radiotherapy on Periodontal and Dental Oral Health: A Prospective Cohort Study
Brief Title: Longitudinal Oral Health Changes After Head and Neck Radiotherapy
Acronym: HN-ORAL-RT
Status: Active, not recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma ElSayed, assistant professor, Ain Shams University
Other Study IDs: HAMO0223
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Head & Neck Cancer; Head & Neck Squamous Cell Carcinoma; Periodontal Disease; Xerostomia
Keywords: Head and neck radiotherapy; periodontal health; radiation-induced oral complications; dental caries; salivary dysfunction; oral health quality of life
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Periodontal Diseases; Xerostomia; Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and Neck Radiotherapy Cohort: Adult patients with head and neck cancer undergoing standard external beam radiotherapy who are followed longitudinally to evaluate periodontal health, dental outcomes, salivary function, and oral health-related quality of life.

SUMMARY:
This prospective observational study evaluates how head and neck radiotherapy affects oral health over time. Patients with head and neck cancer undergoing standard radiotherapy are followed from before treatment through multiple post-treatment visits. Changes in periodontal health, dental status, salivary function, and patient-reported oral health quality of life are assessed. The study aims to better understand the long-term oral complications of radiotherapy and to support improved preventive and supportive dental care for cancer patients.

DETAILED DESCRIPTION:
This prospective longitudinal cohort study investigates the effects of head and neck radiotherapy on periodontal health, dental outcomes, salivary gland function, and oral health-related quality of life.

Adult patients with histologically confirmed head and neck malignancies scheduled to receive external beam radiotherapy are enrolled and followed longitudinally. Clinical assessments are conducted at baseline prior to radiotherapy, at the end of radiotherapy, and at 3, 6, and 12 months post-treatment.

Periodontal evaluation includes clinical attachment level, probing pocket depth, plaque index, gingival index, and bleeding on probing, recorded at six sites per tooth using standardized periodontal examination protocols. Dental outcomes include decayed, missing, and filled teeth index, radiation-associated caries incidence, and tooth mobility. Salivary gland function is assessed using unstimulated whole saliva collection. Patient-reported outcomes include xerostomia severity and oral health-related quality of life using validated questionnaires.

Radiotherapy characteristics including technique, total dose, fractionation schedule, mandibular field involvement, and concurrent chemotherapy are recorded. Longitudinal changes in oral health outcomes are analyzed to identify patterns of disease progression and potential predictors of radiotherapy-related oral complications.

This study aims to generate clinical evidence to improve preventive strategies, early detection, and supportive oral care protocols for patients receiving head and neck radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed head and neck malignancy
* Planned radiotherapy dose ≥50 Gy
* Presence of at least 20 natural teeth
* No periodontal treatment during the preceding 6 months
* Ability to comply with the scheduled follow-up visits

Exclusion Criteria:

* Previous head and neck radiotherapy
* Autoimmune salivary gland disorders
* Current bisphosphonate or anti-resorptive therapy
* Pregnancy
* Uncontrolled systemic disease (HbA1c >9% for diabetic patients)
* Severe periodontal destruction requiring immediate surgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with head and neck cancer receiving external beam radiotherapy at a tertiary referral hospital who are followed longitudinally for oral and periodontal health outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-25 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Attachment Level (CAL) | Baseline, end of radiotherapy, and 3, 6, 9, and 12 months post-radiotherapy
  Mean change in clinical attachment level measured in millimeters using a standardized UNC-15 periodontal probe at six sites per tooth. CAL is used as the primary indicator of periodontal tissue loss following radiotherapy.

SECONDARY OUTCOMES:
Change in Probing Pocket Depth (PPD) | Baseline, end of radiotherapy, and 3, 6, 9, and 12 months post-radiotherapy
  Mean probing pocket depth measured in millimeters at six sites per tooth using a standardized UNC-15 periodontal probe as an indicator of periodontal pocket severity.
Change in Bleeding on Probing (BOP) | Baseline, end of radiotherapy, and 3, 6, 9, and 12 months post-radiotherapy
  Percentage of periodontal sites exhibiting bleeding on probing as a measure of periodontal inflammation.
Change in Decayed, Missing, and Filled Teeth (DMFT) Index | Baseline, end of radiotherapy, and 3, 6, 9, and 12 months post-radiotherapy
  Dental caries experience assessed using the Decayed, Missing, and Filled Teeth (DMFT) index to evaluate cumulative dental disease burden.
Change in Xerostomia Inventory Score | Baseline, end of radiotherapy, and 3, 6, 9, and 12 months post-radiotherapy
  Patient-reported xerostomia severity measured using the validated Xerostomia Inventory questionnaire.
Change in Unstimulated Salivary Flow Rate | Baseline, end of radiotherapy, and 3, 6, 9, and 12 months post-radiotherapy
  Unstimulated whole salivary flow rate measured in milliliters per minute using the passive drooling collection method.
Change in Oral Health Impact Profile-14 (OHIP-14) Score | Baseline, end of radiotherapy, and 3, 6, 9, and 12 months post-radiotherapy
  Oral health-related quality of life assessed using the OHIP-14 questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Maher Teaching Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No